CLINICAL TRIAL: NCT00355563
Title: Use of the PAS-Port Proximal Anastomosis System for Creation of Aorto-Venous Proximal Anastomoses in Coronary Bypass Surgery
Brief Title: Study of the PAS-Port® Proximal Anastomosis System in Coronary Bypass Surgery
Acronym: EPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardica, Inc (Industry)
Responsible Party: Ric Ruedy, Vice President, RA/CA/QA, Cardica, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IP2005-07
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PAS-Port Automated Proximal Anastomosis System

SUMMARY:
The study has been designed to comparatively evaluate the safety and effectiveness of the PAS-Port Proximal Anastomosis System and conventional suturing techniques for creation of the connection between graft veins and the aorta in patients undergoing coronary artery bypass graft surgery for treatment of coronary artery disease. Patients in the study will have a coronary angiogram approximately 9 months following surgery to determine the patency of vein grafts created using either the automated PAS-Port or hand sewn methods. Safety will be evaluated by documenting the occurence of adverse clinical events and evealuating possible association with either method.

ELIGIBILITY:
PRE-OPERATIVELY

Inclusion Criteria:

* Able to give informed consent, able to understand the intent and clinical meaning of the study as well as its implications. Patient is legally competent.
* Assessment that the patient is willing and able to have follow-up visits and examinations
* Age greater than or equal to 50 years and less than 85 years
* Ejection fraction of >30%
* Can tolerate radiographic contrast media
* Requires non-emergent coronary artery bypass with at least two vein bypass grafts intended
* Coronary artery targets intended for bypass index grafts must have >70% native stenosis
* Life expectancy >1 year

Exclusion Criteria:

* Patient is participating in other clinical trials that would conflict with this protocol
* Unable to meet study requirements (travel, general health)
* Pregnancy
* Previous cardiac surgery
* Requiring preoperative use of an intraaortic balloon pump
* Congestive heart failure / NYHA Class IV
* History of thromboembolic disease requiring ongoing anticoagulation therapy or the presence of a bleeding disorder
* Acute or chronic dialysis
* Creatinine of greater than 200 µmol/L (2.3 mg/dL) in the last 30 days
* Documented acute or suspected systemic infection
* Need for ongoing immunosuppressive therapy
* Recent (less than 2 weeks) history of cerebrovascular accident
* Aspirin allergy or other contraindications to aspirin use

INTRA-OPERATIVELY

Inclusion Criteria:

* Patient is hemodynamically stable
* Open chest reassessment of the revascularization strategy confirms that two vein bypass grafts are still intended
* Target vessel wall properties that are suitable for performing both a hand-sewn and a PAS-Port anastomosis
* Target vessel is greater than 1.8 mm in diameter at sites where anastomoses are planned
* Target vessel at sites where anastomoses will be placed are free from severe calcifications or severe atheromas
* The length of the vein graft(s) is adequate for both of the planned index graft revascularization strategies
* Vein outside diameter and double wall thickness are between 4 and 6 mm(inclusive) and less than or equal to 1.4 mm, respectively, at the graft site intended for the PAS-Port proximal anastomosis
* The vein(s) is of suitable quality to be used as a bypass graft conduit

Exclusion Criteria:

-Any of the Intra-operative Inclusion Criteria not met

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Graft Patency at 9 months post-operatively
Safety: Peri-and Post-operative MACE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: John Puskas, M.D., Principal Investigator — Emory University
Locations (1):
- St. Michael's Medical Center, Newark, New Jersey, United States